CLINICAL TRIAL: NCT00071643
Title: Prevention of Post-Stroke Depression - Treatment Strategy
Brief Title: Preventing Post-Stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert G. Robinson (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Robert G. Robinson, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 200207091; R01MH065134 (NIH); DATR A4-GPX
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Depression; Cerebrovascular Accident
Keywords: Stroke
MeSH Terms: conditions — Depression; Stroke | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 Problem Solving Therapy (Experimental): Participants will receive problem solving therapy.
  Interventions: Behavioral: Problem Solving Therapy
- 2. Escitalopram (Experimental): Participants will receive escitalopram.
  Interventions: Drug: Escitalopram
- 3 Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem solving therapy aims to make patients aware of symptoms of problems and link those with behaviors associated with solving them.
  Arms: 1 Problem Solving Therapy
Drug: Escitalopram — Participants will receive escitalopram, a selective serotonin reuptake inhibitor.
  Other Names: Lexapro
  Arms: 2. Escitalopram
Other: Placebo — Participants will receive a placebo pill.
  Arms: 3 Placebo

SUMMARY:
This study will evaluate the effectiveness of both drug and non-drug treatments in preventing depression after a stroke.

DETAILED DESCRIPTION:
The development of depression after a stroke is a serious condition that can have negative effects on thought, emotions, and overall daily functioning, particularly in the first year following the stroke. Evidence suggests that antidepressants may be used to prevent post-stroke depression. This study will treat nondepressed stroke patients with antidepressants or problem solving therapy (PST) to determine the most effective treatments for preventing depression.

Participants in this study will be randomly assigned to receive PST, escitalopram, or placebo (an inactive pill) for 12 months. Participants who display depressive symptoms for 2 weeks or more will be removed from the study. After 12 months, treatment will be discontinued and participants will be monitored for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Stroke within the last 120 days

Exclusion Criteria:

* DSM (Diagnostic and Statistical Manual) IV criteria for major or minor depressive disorder
* Heart, respiratory, kidney, or liver failure; severely disabling musculoskeletal disorder; or cancer
* Diagnosis of neurodegenerative disorders such as Parkinson's disease, Alzheimer's disease, Multiple System Atrophy, or Huntington's disease
* Pre-existing dementia or aphasia with severe language comprehension deficits
* Alcohol or substance abuse or dependence within the last 12 months
* Recurrent unipolar or bipolar disorder prior to the stroke

Ages: 31 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2002-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Incidence of depressive disorders in the study population | Measured at baseline, Week 6, and Months 3, 6, 9, 12, and 18

SECONDARY OUTCOMES:
Functional Independence Measure | Measured at baseline, at Week 6, and at Months 3, 6, 9, 12, and 18
Stroke Impact Scale | Measured at baseline, Week 6, and Months 3, 6, 9, 12, and 18
Neurocognitive tests of executive functions and speed of information processing | Measured at baseline and after 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Burke Rehabilitation Hospital, White Plains, New York

REFERENCES:
- [Derived] Mikami K, Jorge RE, Moser DJ, Arndt S, Jang M, Solodkin A, Small SL, Fonzetti P, Hegel MT, Robinson RG. Increased frequency of first-episode poststroke depression after discontinuation of escitalopram. Stroke. 2011 Nov;42(11):3281-3. doi: 10.1161/STROKEAHA.111.626507. Epub 2011 Aug 25. PMID 21868736
- [Derived] Jorge RE, Acion L, Moser D, Adams HP Jr, Robinson RG. Escitalopram and enhancement of cognitive recovery following stroke. Arch Gen Psychiatry. 2010 Feb;67(2):187-96. doi: 10.1001/archgenpsychiatry.2009.185. PMID 20124118
- [Derived] Robinson RG, Jorge RE, Moser DJ, Acion L, Solodkin A, Small SL, Fonzetti P, Hegel M, Arndt S. Escitalopram and problem-solving therapy for prevention of poststroke depression: a randomized controlled trial. JAMA. 2008 May 28;299(20):2391-400. doi: 10.1001/jama.299.20.2391. PMID 18505948